CLINICAL TRIAL: NCT01916200
Title: Efficacy and Safety of Paroxetine Controlled Release for Major Depressive Disorder in Irritable Bowel Syndrome Patients: An Open-label, Randomized, add-on Study
Brief Title: Efficacy and Safety of Paroxetine Controlled Release for Major Depressive Disorder in Irritable Bowel Syndrome Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was Cancelled Before Active
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117049
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine CR group (Experimental): Paroxetine CR plus IBS regular treatment group
  Interventions: Drug: Paroxetine CR
- Blank group (No Intervention): IBS regular treatment group

INTERVENTIONS:
Drug: Paroxetine CR — Paroxetine CR will be provided by GlaxoSmithKline (GSK) and be available as 12.5 mg over-encapsulated tablets with the research use only label outside the package. Paroxetine CR should be administered as a single daily dose, with or without food. The recommended initial dose is 25 mg/day. Patients were dosed in a range of 25 mg to 62.5 mg/day in the clinical trials demonstrating the effectiveness of paroxetine CR in the treatment of major depressive disorder. As with all drugs effective in the treatment of major depressive disorder, the full effect may be delayed. Some patients not responding to a 25-mg dose may benefit from dose increases, in 12.5 mg/day increments, up to a maximum of 62.5 mg/day. Dose changes should occur at intervals of at least 1 week.
  Arms: Paroxetine CR group

SUMMARY:
This is an open label, randomized, add-on, 8 weeks multicentre study to evaluate the efficacy and safety of paroxetine Controlled Release (CR) in patients with Major Depressive Disorder (MDD) comorbid Irritable Bowel Syndrome (IBS).

Subjects will be patients who are referred to the outpatient or inpatient clinic of gastroenterology departments of province level general hospitals in China. All subjects present with irritable bowel syndrome according to ROME III, and also are diagnosed with MDD by Mini-International Neuropsychiatric Interview (MINI). All subjects will provide written informed consent prior to participating in the study. Subjects will be assessed for eligibility at a screening visit, with eligible patients returning for a assessment within 1 week, at which time they will randomly enter into paroxetine CR (12.5mg/d, flexible dose: 12.5-50mg/d) plus IBS regular treatment or IBS regular treatment only. Subjects will be evaluated at weeks 2 (Day 14), 4 (Day 28), 6 (Day 42) and 8 (Day 56), for a total of 5 study treatment visits.

DETAILED DESCRIPTION:
This is an open label, randomized, add-on, 8 weeks multicentre study to evaluate the efficacy and safety of paroxetine CR in patients with MDD comorbid IBS.

This study is designed with a 1-week screening period, followed by 8 weeks of treatment and 1 week follow up period, 7 visits totally; the calculation of visit date is base on the real date of random date.

Study Screening:

Visit 1: a screening period for within 7 days to determine eligibility for the study, subjects aged ≥ 18 and ≤ 65 years at the time of screening, must have a diagnosis of IBS and MDD. After giving their informed consent to participate in the study, patients will undergo screening assessments, including demographic data (birth, race, gender, height, weight), medical history, disease history, therapy history, concomitant medication, physical examination, vital signs, 12-lead ECG and laboratory assessments.

Treatment Phase:

The treatment phase will last for 8 weeks. The visit (except baseline) will have ±3 days.

Visit 2 (Day 0, baseline visit): Patients who fulfil all the study inclusion and exclusion criteria will accept baseline assessment (including concomitant medication, vital signs and scale assessment) and be randomised into paroxetine CR plus IBS regular treatment group or IBS regular treatment only group at baseline visit. The day after randomizing (Day 1), patients will receive paroxetine CR 12.5mg/d plus IBS regular treatment or IBS regular treatment only (patients who have received IBS regular treatment before can continue their treatment). On Day 8, following 1 weeks of treatment, paroxetine CR should be titrated to 25mg/d.

Visit 3-5 (Day 14, Day 28, Day 42): Efficacy and safety assessments will be performed at these visits, including vital signs and HDRS-17 (Hamilton Depression Rating Scale 17 items), CGI-S (Clinical Global Impression- Severity), CGI-I (Clinical Global Impression- Improvement), WHOQOL (World Health Organization Quality of Life Assessment), IBSSS (The Irritable Bowel Severity Scoring System). From Week 3 to 6, the investigator can titrate the subject's dose upwards according to clinical response and tolerability, at a maximum rate of paroxetine CR 12.5mg every 14 days. For example, if CGI-I is ≥3 based on the assessment at scheduled clinic visit, and the patient is able to tolerate an increased dose, the dose increment to the next dose level shall be considered. The highest dose that may be administered is paroxetine CR 50 mg and dose titration may only occur at scheduled visits.

Visit 6 (Day 56): Efficacy and safety assessments will be performed at these visits, including vital signs, physical examination, laboratory assessments and HDRS-17, CGI-S, CGI-I, WHOQOL, IBSSS.

If the patient experiences an adverse event (AE) and the investigator deems that a reduction in dose is required then the patient may be administered a dose one level (paroxetine CR 12.5 mg) lower than they were taking previously. Upon resolution of the AE, the investigator may return to patient's pre-AE dose level.

Follow-Up:

After treatment phase, the investigator should communicate with all the subjects about the follow-up choice: reduce or continuing paroxetine CR treatment/ other antidepressants treatment/ transferring to psychiatric clinics. It is not recommend to reduce drug dosage during the treatment period of MDD.

For those subjects who decide to discontinue paroxetine CR treatment: a gradual reduction in the dose rather than abrupt cessation is recommended whenever possible. The dosage should be reduced weekly, the daily dose reduction is 12.5mg per week, and once a week. If intolerable symptoms occur following a decrease in the dose or upon discontinuation of treatment, then resuming the previously prescribed dose may be considered. Subsequently, the physician may continue decreasing the dose but at a more gradual rate.

Visit 7 (Day 63): the investigator should conduct safety follow up by phone call to all participants to investigate the medication situation and safety related information.

Withdraw:

Patients withdrawn from the study prior to Visit 6 (Week 8) will have all end-of-study procedures performed. Patients withdrawn from the study for any reason are to attend an early withdrawal visit on withdrawal from the study. In addition, patients have to taper the study drug if they end the study on a dose level higher than dose level 1 (paroxetine CR 12.5 mg). The dosage should be reduced weekly, the daily dose reduction is 12.5mg per week, and once a week.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic for IBS according to ROME III;
2. Meet the diagnostic for MDD according to MINI;
3. Age≥18 and ≤ 65;
4. Patients or their guardian have the ability to understand and to provide informed consent to the examination, observation, and evaluation; processes specified in this protocol, and have signed the informed consent from based on a full understanding of the trial.

Exclusion Criteria:

1. Patients were also excluded if they had any medical condition that would contraindicate the use of paroxetine CR [Seroxat CR®];
2. History of alcohol / drug dependence and schizophrenia; history of serious mental illness;
3. Major neurological deficits that interfere with the patient's ability to understand the study procedures and provide a written informed consent;
4. Patients were also excluded if their current episode of depression had failed to respond to two or more adequate trials of antidepressants, benzodiazepines, or other anxiolytics at a clinically appropriate dose for a minimum of 4 weeks;
5. Suicide ideation;
6. Use monoamine oxidase inhibitors (MAOIs), benzodiazepines or other antidepressants within at least 14 days before study begin;
7. Other medical and psychological conditions prevent patients from participating in the study or signing informed consent;
8. Pregnant or lactating females, or anyone who plan to become pregnant during the study period;
9. Those who are known to currently participate a clinical trial;
10. Those patients with significant organ disease. GI disorders that are infectious;
11. Ischemic, radiation-induced, or medication-induced; inflammatory bowel disease (Cohn's disease and ulcerative colitis);
12. Recent gastrointestinal surgery (within 6 months).
13. Has received electroconvulsive therapy (ECT) or psychotherapy in the 3 months prior to screening.
14. Presents with clinically significant abnormalities in haematology, clinical chemistry, electrocardiogram (ECG) or physical examination at screening which have not resolved prior to the baseline visit or has clinically significant conditions, which in the opinion of the investigator, will render the patient unsuitable for the study and pose a safety concern or interfere with the accurate safety and efficacy assessments (e.g., severe cardiovascular disease, hepatic or renal failure etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
HDRS-17 | 8 weeks

SECONDARY OUTCOMES:
HDRS-17 item 10 | 8 weeks
CGI-I | 8 weeks
CGI-S | 8 weeks
WHOQOL | 8 weeks
IBSSS | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Mertz HR. Irritable bowel syndrome. N Engl J Med. 2003 Nov 27;349(22):2136-46. doi: 10.1056/NEJMra035579. No abstract available. PMID 14645642
- [Background] Creed F, Fernandes L, Guthrie E, Palmer S, Ratcliffe J, Read N, Rigby C, Thompson D, Tomenson B; North of England IBS Research Group. The cost-effectiveness of psychotherapy and paroxetine for severe irritable bowel syndrome. Gastroenterology. 2003 Feb;124(2):303-17. doi: 10.1053/gast.2003.50055. PMID 12557136
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] Cho HS, Park JM, Lim CH, Cho YK, Lee IS, Kim SW, Choi MG, Chung IS, Chung YK. Anxiety, depression and quality of life in patients with irritable bowel syndrome. Gut Liver. 2011 Mar;5(1):29-36. doi: 10.5009/gnl.2011.5.1.29. Epub 2011 Mar 16. PMID 21461069
- [Background] Drossman DA, Li Z, Andruzzi E, Temple RD, Talley NJ, Thompson WG, Whitehead WE, Janssens J, Funch-Jensen P, Corazziari E, et al. U.S. householder survey of functional gastrointestinal disorders. Prevalence, sociodemography, and health impact. Dig Dis Sci. 1993 Sep;38(9):1569-80. doi: 10.1007/BF01303162. PMID 8359066
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Russo MW, Gaynes BN, Drossman DA. A national survey of practice patterns of gastroenterologists with comparison to the past two decades. J Clin Gastroenterol. 1999 Dec;29(4):339-43. doi: 10.1097/00004836-199912000-00009. PMID 10599638
- [Background] Gros DF, Antony MM, McCabe RE, Swinson RP. Frequency and severity of the symptoms of irritable bowel syndrome across the anxiety disorders and depression. J Anxiety Disord. 2009 Mar;23(2):290-6. doi: 10.1016/j.janxdis.2008.08.004. Epub 2008 Aug 27. PMID 18819774
- [Background] Sandler RS. Epidemiology of irritable bowel syndrome in the United States. Gastroenterology. 1990 Aug;99(2):409-15. doi: 10.1016/0016-5085(90)91023-y. PMID 2365191
- [Background] Boyce PM, Talley NJ, Balaam B, Koloski NA, Truman G. A randomized controlled trial of cognitive behavior therapy, relaxation training, and routine clinical care for the irritable bowel syndrome. Am J Gastroenterol. 2003 Oct;98(10):2209-18. doi: 10.1111/j.1572-0241.2003.07716.x. PMID 14572570
- [Background] Guthrie E, Creed F, Fernandes L, Ratcliffe J, Van Der Jagt J, Martin J, Howlett S, Read N, Barlow J, Thompson D, Tomenson B. Cluster analysis of symptoms and health seeking behaviour differentiates subgroups of patients with severe irritable bowel syndrome. Gut. 2003 Nov;52(11):1616-22. doi: 10.1136/gut.52.11.1616. PMID 14570732
- [Background] Masand PS, Kaplan DS, Gupta S, Bhandary AN, Nasra GS, Kline MD, Margo KL. Major depression and irritable bowel syndrome: is there a relationship? J Clin Psychiatry. 1995 Aug;56(8):363-7. PMID 7635853
- [Background] Vandvik PO, Lydersen S, Farup PG. Prevalence, comorbidity and impact of irritable bowel syndrome in Norway. Scand J Gastroenterol. 2006 Jun;41(6):650-6. doi: 10.1080/00365520500442542. PMID 16716962
- [Background] Park JM, Choi MG, Cho YK, Lee IS, Kim JI, Kim SW, Chung IS. Functional Gastrointestinal Disorders Diagnosed by Rome III Questionnaire in Korea. J Neurogastroenterol Motil. 2011 Jul;17(3):279-86. doi: 10.5056/jnm.2011.17.3.279. Epub 2011 Jul 13. PMID 21860820
- [Background] Cremonini F, Talley NJ. Irritable bowel syndrome: epidemiology, natural history, health care seeking and emerging risk factors. Gastroenterol Clin North Am. 2005 Jun;34(2):189-204. doi: 10.1016/j.gtc.2005.02.008. PMID 15862929
- [Background] Hillila MT, Siivola MT, Farkkila MA. Comorbidity and use of health-care services among irritable bowel syndrome sufferers. Scand J Gastroenterol. 2007 Jul;42(7):799-806. doi: 10.1080/00365520601113927. PMID 17558902
- [Background] Friedrich M, Grady SE, Wall GC. Effects of antidepressants in patients with irritable bowel syndrome and comorbid depression. Clin Ther. 2010 Jul;32(7):1221-33. doi: 10.1016/j.clinthera.2010.07.002. PMID 20678672
- [Background] Creed F, Ratcliffe J, Fernandez L, Tomenson B, Palmer S, Rigby C, Guthrie E, Read N, Thompson D. Health-related quality of life and health care costs in severe, refractory irritable bowel syndrome. Ann Intern Med. 2001 May 1;134(9 Pt 2):860-8. doi: 10.7326/0003-4819-134-9_part_2-200105011-00010. PMID 11346322
- [Background] Thompson W, Longstreth G, Drossman Deds. Functional bowel disorders and functional abdominal pain. In: Drossman DA, Corazziari E, Talley NJ, Thompson WG, Whitehead WE, eds. Rome II. The Functional Gastrointestinal Disorders, 2nd edn. McLean, VA: Degnon Associates, 2000: 351-432.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Background] Mitchell CM, Drossman DA. Survey of the AGA membership relating to patients with functional gastrointestinal disorders. Gastroenterology. 1987 May;92(5 Pt 1):1282-4. doi: 10.1016/s0016-5085(87)91099-7. No abstract available. PMID 3557021